CLINICAL TRIAL: NCT01485640
Title: A Long-term, Multicenter, Open-Label, Flexible Dose Continuation Study in Subjects Who Have Completed a Prior Lurasidone Study
Brief Title: Lurasidone Extended Use Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1050298; 2011-000682-12 (EudraCT Number)
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Schizophrenia; bipolar disorder; Lurasidone; Latuda
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lurasidone (Experimental): Lurasidone flexibly dosed
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — Lurasidone flexibly dosed; doses of 20, 40, 60 or 80 mg/day will be taken orally with food

SUMMARY:
This is an open-label continuation study designed to monitor the safety, tolerability and effectiveness of lurasidone in subjects who have completed participation in a lurasidone extension study (NCT00868959 and NCT01566162) and who may benefit from continued treatment with lurasidone.

ELIGIBILITY:
Inclusion Criteria:

* The subject or legal guardian provides written informed consent. For eligible subjects under age 18, verbal assent is also required.
* The subject has completed the extension phase of a prior lurasidone clinical study. Eligible subjects may enroll into this continuation study directly (or within 10 days) after completing the extension phase of a prior lurasidone clinical study. Subjects that have completed an extension study prior to the initiation of this protocol at the study site, may participate in this study up to 3 months after completion of the extension phase of the prior lurasidone study.
* The subject is judged by the Investigator to be suitable for participation in a clinical study involving open-label lurasidone treatment and is able to comply with the protocol.
* The subject, in the Investigator's judgment, may benefit from continued treatment with lurasidone

Exclusion Criteria:

* The subject is considered by the Investigator, to be at imminent risk for homicidal or suicidal behavior.
* The subject resides in a country where lurasidone has been approved for any indication.
* The subject is currently enrolled in any other investigational study.
* The subject answers "yes" to "Suicidal Ideation" Items 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (46):
- Okanagan Clinical Trials, Kelowna, British Columbia, Canada
- Colombia (3):
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA Investigations, Barranquilla
  - E.S.E. Hospital Mental de Antioquia, Bello
  - CISNE - UIC Campo Abierto, Bogotá
- Czechia (5):
  - Psychiatricka ambulance, Brno-mesto
  - Vojenska nemocnice Olomouc, Olomouc
  - Clintrial, s.r.o., Prague
  - Psychiatry Trial s.r.o., Prague
  - Medical Services Prague s.r.o., Prague
- France (2):
  - Zans Ritter, Marcel, Orvault
  - Hôpital Chalucet, Centre hospitalier intercommunal de Toulon la Seyne sur mer (CHITS), Toulun
- India (11):
  - Brain Mind Behavior Neuroscience Research Institute, Visakhapatnam, Andh Prad
  - Vijayawada Institute of Mental Health and Neurosciences, Vijayawada, Andhra Pradesh
  - Samvedna Hospitals, Ahmedabad, Gujarat
  - Seth K M School of P G Medicine & Research, Ahmedabad, Gujarat
  - Mental Health Treatment Rehabililitation Foundation Dept. of Psychiatry, Ahmedabad, Gujarat
  - Hatkesh Healthcare Foundation, Jūnāgadh, Gujarat
  - Brij Psychiatry Hospital & Muskaan Research Centre, Vadodara, Gujarat
  - Shanti Nursing Home, Aurangabad, Maharashtra
  - Dr. Tambi's Neuropsychiatry Center, Jaipur, Rajaasthan
  - R.K. Yadav Memorial Mental Health & De-Addiction Hospital Psychiatry, Jaipur, Rajasthan
  - Mahendru Psychiatric Centre, Kanpur
- Lithuania (3):
  - Neuromeda JSC, Kaunas
  - JSC Neuromeda, Kaunas
  - Seskines Outpatient Clinic, Public Institution, Vilnius
- Romania (2):
  - Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca
  - Spitalul Clinic de Neuropsihiatrie Craiova, Craiova
- Russia (4):
  - Regional Government Institution (RGI) 'Lipetsk Regional Psychoneurology Hospital', Lipetsk
  - St. Petersburg State Budgetary Healthcare Institution 'City Psychoneurology Dispensary #7 (with In-Patient Department)', (SPb SBHI "CPNDD-7"), at Daycare Facility #1, Saint Petersburg
  - St. Petersburg State Government Healthcare Institution "City Psychiatric Hospital #4" (St. Petersburg Insane Asylum Distributor), Saint Petersburg
  - St. Petersburg State Healthcare Institution (SPbSHI) "City Psychiatric Hospital #6", Saint Petersburg
- Serbia (2):
  - Institute of Mental Health, Belgrade
  - Clinical Centre Nis, Clinic for mental health protection, Niš
- Slovakia (4):
  - Psychiatricka ambulancia Mentum s.r.o., Bratislava
  - PsychoLine s.r.o. Psychiatricka ambulancia, Rimavská Sobota
  - Centrum zdravia R.B.K. s.r.o. Psychiatricka ambulancia, Svidník
  - Pro mente sana s.r.o. Psychiaricka ambulancia, Trenčín
- South Africa (3):
  - Dey Clinic, Pretoria, Gauteng
  - Cape Trial Centre, Tygervalley, Western Cape
  - Denmar Hospital Consulting Rooms, Pretoria
- Ukraine (6):
  - Kherson Regional Psychiatric Hospital, Kherson, Vil Stepanivka
  - Dnipropetrovsk Regional Clinical Hospital named Mechnikov, Dnipropetrovsk
  - Regional Clinical Psychiatric Hospital, Dept #11, Donetsk
  - Institute of Neurology, Psychiatry and Narcology, NAMS of Ukraine, Khardov
  - Crimean republican Clinical Psychiatric Hospital, Simferopol
  - Reg. Psych. Hosp.n.a.O.Yuschenko, Dept #21, Vinnitsia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lurasidone
Started | 162
Completed | 40
Not Completed | 122
Not completed — Adverse Event | 10
Not completed — Lack of Efficacy | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 14
Not completed — Terminated by Sponsor | 95

BASELINE CHARACTERISTICS:
Arm/Group | Lurasidone
Number analyzed (Participants) | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 159
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 32
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 105
  More than one race | 0
  Unknown or Not Reported | 20
Region of Enrollment [Number; unit: participants]
  Serbia | 6
  France | 6
  Czech Republic | 25
  Slovakia | 17
  Canada | 3
  Ukraine | 11
  Romania | 2
  Lithuania | 8
  Russian Federation | 20
  South Africa | 26
  Colombia | 6
  India | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent AEs, SAEs or Who Discontinued Due to AEs
Description: Primary Safety assessments included spontaneous adverse event (AE) and serious adverse events (SAEs) monitoring.
Time Frame: 18 months
Population: Safety Population - subjects who took at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Lurasidone
Number analyzed (Participants) | 162
participants
  Subject with at least on treatment emergent AE | 63
  Subject with at least one treatment emergent SAE | 7
  Subjects discontinued due to TEAE | 10

2. Secondary Outcome: Change From Baseline to Month 18 (LOCF) in the Clinical Global Impression Severity Score (CGI-S
Description: The CGI-S score is a single value, clinician-rated assessment of illness severity and ranges from 1= 'Normal, not at all ill' to 7= 'Among the most extremely ill patients'. A higher score is associated with greater illness severity.
Time Frame: 18 months
Population: Only 153 subjects who had baseline and at least one post-baseline assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 153
units on a scale | -0.18 (0.877)

ADVERSE EVENTS:
Time Frame: 18 Months
Arm/Group | Lurasidone
Serious Adverse Events (participants affected / at risk) | 7/162
Other Adverse Events (participants affected / at risk) | 40/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=162)
Pilonidal cyst (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Depression suicidal (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 2 (2)
Schizophrenia, paranoid type (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=162)
Diarrhoea (Gastrointestinal disorders) | 6 (8)
Vomiting (Gastrointestinal disorders) | 5 (11)
Nausea (Gastrointestinal disorders) | 4 (4)
Influenza (Infections and infestations) | 6 (6)
Nasopharyngitis (Infections and infestations) | 6 (9)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4)
Hepatic enzyme increase (Investigations) | 4 (4)
Headache (Nervous system disorders) | 9 (12)
Anxiety (Psychiatric disorders) | 5 (11)
Insomnia (Psychiatric disorders) | 5 (6)
Depression (Psychiatric disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS agreement between Principal Investigator and Sponsor that restricts PI's rights to discuss or publish trial results after trial is completed.

In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication provided, if a multicenter publication is not forthcoming within 24 months post completion of study at all sites, PI shall be free to publish.